CLINICAL TRIAL: NCT03685773
Title: The Role of Hepatic Denervation in the Dysregulation of Glucose Metabolism in Liver Transplant Recipients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Permanently terminated due to COVID-19 given the poor vaccine penetrance in liver transplant recipients.
  This is not a suspension of IRB approval.
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018-9506
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2; Glucose, High Blood; Glucose Metabolism Disorders
Keywords: diabetes; type 2 diabetes; diazoxide; insulin resistance; MRI; liver transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Diabetes Mellitus; Insulin Resistance | interventions — Diazoxide; Niacin

STUDY DESIGN:
Who Masked: Participant
Masking Description: The subject will be blinded to which study drug is received first (Drug or Placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- MRI: Non-diabetic transplant (Diazoxide) (Experimental): Diazoxide (up to 7 mg/kg)
  Interventions: Drug: Diazoxide
- MRI: Non-diabetic transplant (Placebo) (Placebo Comparator): Taste-matched placebo for diazoxide
  Interventions: Drug: Placebo (for diazoxide)
- MRI: T2D transplant (Diazoxide) (Experimental): Diazoxide (up to 7 mg/kg)
  Interventions: Drug: Diazoxide
- MRI: T2D transplant (Placebo) (Placebo Comparator): Taste-matched placebo for diazoxide
  Interventions: Drug: Placebo (for diazoxide)
- Clamp: Non-diabetic transplant (Diazoxide) (Experimental): Diazoxide (up to 7 mg/kg) before pancreatic clamp study
  Interventions: Drug: Diazoxide
- Clamp: Non-diabetic transplant (Placebo) (Placebo Comparator): Taste-matched placebo (for diazoxide) before pancreatic clamp study
  Interventions: Drug: Placebo (for diazoxide)
- Clamp: T2D transplant (Diazoxide) (Experimental): Diazoxide (up to 7 mg/kg) before pancreatic clamp study
  Interventions: Drug: Diazoxide
- Clamp: T2D transplant (Placebo) (Placebo Comparator): Taste-matched placebo (for diazoxide) before pancreatic clamp study
  Interventions: Drug: Placebo (for diazoxide)
- Clamp: T2D transplant (Diazoxide + Nicotinic Acid) (Experimental): Nicotinic acid infusion and diazoxide (up to 7 mg/kg) before pancreatic clamp study
  Interventions: Drug: Diazoxide; Drug: Nicotinic acid
- Clamp: T2D transplant (Placebo + Nicotinic Acid) (Experimental): Nicotinic acid infusion and placebo (for diazoxide) before pancreatic clamp study
  Interventions: Drug: Placebo (for diazoxide); Drug: Nicotinic acid
- MRI: T2D transplant (Diazoxide + Nicotinic Acid) (Experimental): Nicotinic acid infusion and diazoxide (up to 7 mg/kg)
  Interventions: Drug: Diazoxide; Drug: Nicotinic acid
- MRI: T2D transplant (Placebo + Nicotinic Acid) (Experimental): Nicotinic acid infusion and placebo (for diazoxide)
  Interventions: Drug: Placebo (for diazoxide); Drug: Nicotinic acid

INTERVENTIONS:
Drug: Diazoxide — MRI studies: Non-diabetic and T2D participants will receive diazoxide (up to 7 mg/kg) between baseline MRI scan and second MRI scan.
  Clamp studies: Non-diabetic participants will not require an overnight admission. They will receive diazoxide (up to 7 mg/kg) and undergo the pancreatic clamp study. Type 2 diabetic participants will be admitted the evening before the study day to normalize blood sugar levels. They will then receive diazoxide (up to 7 mg/kg) the next morning and undergo the pancreatic clamp study.
  Other Names: Proglycem
  Arms: Clamp: Non-diabetic transplant (Diazoxide); Clamp: T2D transplant (Diazoxide + Nicotinic Acid); Clamp: T2D transplant (Diazoxide); MRI: Non-diabetic transplant (Diazoxide); MRI: T2D transplant (Diazoxide + Nicotinic Acid); MRI: T2D transplant (Diazoxide)
Drug: Placebo (for diazoxide) — MRI studies: Non-diabetic and T2D participants will receive placebo (for diazoxide) between baseline MRI scan and second MRI scan.
  Clamp studies: Non-diabetic participants will not require an overnight admission. They will receive a taste-matched placebo (for diazoxide) and undergo the pancreatic clamp study. Type 2 diabetic participants will be admitted the evening before the study day to normalize blood sugar levels. They will then receive a taste-matched placebo (for diazoxide) the next morning and undergo the pancreatic clamp study.
  Other Names: Placebo
  Arms: Clamp: Non-diabetic transplant (Placebo); Clamp: T2D transplant (Placebo + Nicotinic Acid); Clamp: T2D transplant (Placebo); MRI: Non-diabetic transplant (Placebo); MRI: T2D transplant (Placebo + Nicotinic Acid); MRI: T2D transplant (Placebo)
Drug: Nicotinic acid — Type 2 diabetic participants in this arm will receive a nicotinic acid infusion to lower free fatty acid levels. They will then receive diazoxide (up to 7 mg/kg) the next morning and undergo the MRI or pancreatic clamp study.
  Other Names: Niacin
  Arms: Clamp: T2D transplant (Diazoxide + Nicotinic Acid); Clamp: T2D transplant (Placebo + Nicotinic Acid); MRI: T2D transplant (Diazoxide + Nicotinic Acid); MRI: T2D transplant (Placebo + Nicotinic Acid)

SUMMARY:
It is believed that important brain centers send signals through the vagus nerve to the liver to suppress the amount of glucose (sugar) that gets produced. People who have received liver transplants have had their vagus nerve cut during transplantation, and many of these individuals have diabetes at one year post-transplant. The goals of this study are: to see whether metabolic control centers in the brain can still be activated normally with the medication diazoxide in patients who have had a liver transplant, and to understand whether disrupting the vagus nerve would result in excess glucose being produced by the liver (ie. a potential mechanism for why these patients develop diabetes).

DETAILED DESCRIPTION:
In this study, investigators will study both diabetic and non-diabetic individuals who are otherwise healthy more than one year after receiving a liver transplant. They will participate in at least one of the following two parts of this study: The first involves functional magnetic resonance imaging (fMRI), and the second is using a day-long infusion study called a "pancreatic clamp."

Functional magnetic resonance imaging (fMRI) is a technique for measuring and mapping brain activity that is noninvasive and safe. This technique relies on the fact that blood flow in the brain and the activity of brain cells are coupled. Investigators will observe the activity of metabolically-relevant areas of the brain by activating potassium channels with diazoxide at baseline and at 2-hour intervals vs when given placebo.

In the pancreatic clamp study, glucose (a sugar) and insulin (a hormone produced in the pancreas that regulates the amount of sugar in the blood) are infused with an intravenous catheter. Blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body which are related to glucose metabolism. The rates of endogenous glucose production (a measure of the body's production of sugar) will be measured as the main measurement of the study.

All participants will be screened prior to study enrollment. For the fMRI studies, eligible participants will come on two separate occasions for day-long study visits (one day in which the brain will be imaged before and after receiving diazoxide (a potassium channel activator), and one day in which the brain will be imaged before and after placebo. For the pancreatic clamp studies, eligible participants will come on two separate occasions for day-long study visits (one study with diazoxide, and one study with placebo). All studies in participants with type 2 diabetes will include overnight admissions prior to the study day for gradual normalizing of blood glucose through the infusion of insulin. Participants without diabetes will not have to stay for an overnight admission. Study participants with type 2 diabetes will also be eligible for an additional study in which Nicotinic Acid will be infused overnight to lower free fatty acid (FFA) levels. It will be determined whether FFA lowering will impact the fMRI studies and clamp studies that will be performed the next day.

ELIGIBILITY:
Inclusion Criteria:

* Liver Transplant at least one year ago
* Age: 21-70

Exclusion Criteria:

* BP > 150/90 or <90/60 on more than one occasion, unless there is a documented history of white coat hypertension by treating physician.
* Triglycerides > 400 mg/dl and/or Total Cholesterol >300 mg/dl
* Clinically significant liver dysfunction
* Clinically significant kidney dysfunction, GFR: <60 mg/dL
* Anemia: HgB <12.5 for men and <11.0 for women
* Positive urine drug test. Occasional use of cannabis (once or twice per week) will not be a basis for exclusion.
* Urinalysis: Clinically significant abnormalities
* Clinically significant electrolyte abnormalities
* Smoking >10 cig/day
* Alcohol: Men >14 drinks/wk or >4 drinks/day, Women >7 drinks/wk or >3 drinks/day
* History of active hepatitis infection, HIV/AIDS, chronic kidney disease (stage 3 or greater), active cancer, cardiovascular disease or other heart disease, systemic rheumatologic conditions, seizures, bleeding disorders, muscle disease
* Surgeries that involve removal of endocrine glands except for thyroidectomy (if euthyroid on thyroid hormone replacement - if such history T4 and TSH will be checked)
* Pregnant women
* Subject enrolled in another study less than one month prior to the anticipated start date in the proposed study, besides those done by our group
* Family history: family history of premature cardiac death
* Allergies to medication administered during study
* Uncontrolled psychiatric disorders
* Any condition which in the opinion of the PI makes the subject ill-suited for participation in the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-21 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Endogenous glucose production (EGP) | 7-7.5 hours
  Rates of EGP (a measure of the body's production of sugar) will be measured during pancreatic clamp studies, with suppression of pancreatic hormones by somatostatin infusion and basal hormone replacement.

SECONDARY OUTCOMES:
Change in Arterial Spin Labeling (ASL) signal | Baseline, 2 hours post dosing, 4 hours post dosing
  Change in Arterial Spin Labeling (ASL) signal measured using 3T MRI from baseline to 2 hours post dosing, and 2 hours post dosing to 4 hours post dosing. ASL is a measure of brain blood flow, and an increase in ASL is interpreted as an increase in brain activity. Data is collected at three time points during each of the two visits (pre dosing, 2 hours post dosing, 4 hours post dosing). Response to diazoxide is compared between 3 time points for each group, and this response is then compared between non-diabetic and type 2 diabetic liver transplant subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Hawkins, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States